CLINICAL TRIAL: NCT01311076
Title: A Phase 1, Randomized, Placebo- and Active-Controlled, 4-Period Crossover, Proof of Concept Glucose Clamp Study to Compare the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Properties of Single Doses of TAK-329 With a Single Dose of a Subcutaneously-Injected Rapid-Acting Insulin Analog in Subjects With Type 1 Diabetes Mellitus.
Brief Title: TAK-329 Glucose Clamp Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: TAK-329_102; U1111-1119-7141 (Registry Identifier: WHO)
Record Dates: First submitted 2011-03-07; First posted 2011-03-09 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus; Insulin; Glucose; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Insulin; Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- TAK-329 50 mg (Experimental)
  Interventions: Drug: TAK-329
- TAK-329 200 mg (Experimental)
  Interventions: Drug: TAK-329
- Insulin 0.2 U/kg (Active Comparator)
  Interventions: Drug: Insulin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-329 — TAK-329 50 mg, tablets, orally, single dose, one day.
  Arms: TAK-329 50 mg
Drug: TAK-329 — TAK-329 200 mg, tablets, orally, single dose, one day.
  Arms: TAK-329 200 mg
Drug: Insulin — Insulin 0.2 U/kg, subcutaneous injection, single dose, one day.
  Other Names: Insulin lispro; Humalog
  Arms: Insulin 0.2 U/kg
Drug: Placebo — TAK-329 placebo-matching tablets, orally, single dose, one day.
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the safety, tolerability, pharmacokinetic and pharmacodynamic properties of single doses of TAK-329 with a single dose of a subcutaneously-injected rapid-acting insulin analog in participants with type 1 diabetes mellitus.

DETAILED DESCRIPTION:
Type 1 diabetes mellitus (T1DM), also known as insulin-dependent diabetes mellitus or juvenile-onset diabetes, occurs primarily due to β-cell destruction, usually leading to absolute insulin deficiency. The condition is immune-mediated and is usually idiopathic. Tight glycemic control using intensive insulin therapy was shown in the Diabetes Control and Complications Trial (DCCT) to reduce rates of microvascular complications in T1DM; however, achieving and maintaining such control in T1DM using standard insulin therapy requires a high level of support and is associated with increased potential for hypoglycemia, increased weight gain and, in some patients, aggravation of cardiovascular risk factors including dyslipidemia.

TAK-329 is being developed by Takeda Global Research & Development Center, Inc. (TGRD) as an adjunct treatment to improve glycemic control in patients with type 1 diabetes mellitus who use insulin therapy.

This study will take place at 1 site in the United States. A total of 36 male and female adult participants with T1DM will take part in the study.

The study will last about 77 days, including a 28 days screening period, 4 cross-over treatment periods and a follow up period. Participants will be confined to the study clinic for 2 days in each period. Participants will also be contacted by phone 30 days following the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant or legal guardian is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Is an adult female or an adult male with Type 1 Diabetes Mellitus (diagnosed at least 1 year prior to Screening) with a glycosylated hemoglobin ≤10.0%.
4. Is aged 18 to 50 years, inclusive, at the time of informed consent and first dose of study drug.
5. Weighs at least 50 kg and has a body mass index between 18.0 and 32.0 kg/m2, inclusive at Screening.
6. Males who are nonsterilized and sexually active with a female partner of childbearing potential agree to use adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after the last dose.
7. A female participant, including women of childbearing potential, who is sexually active with a nonsterilized male partner agree to use consistently use contraception from signing of informed consent throughout the duration of the study.
8. Was treated with insulin either in the form of multiple daily injections or as continuous subcutaneous insulin infusion (CSII or "insulin pump") for at least 3 months prior to Screening.
9. Has a fasting serum C-peptide ≤0.2 nmol/L at Screening.
10. The participant, if taking concomitant medications for stable disease, has been on a stable dose for a minimum of 60 days prior to Day 1 of Period 1 and the medications are approved by the investigator and the Takeda Medical Monitor.
11. A female participant of child-bearing potential, if using hormonal contraception, has been on stable hormonal contraception (without changes to the dose or type of preparation) for at least 6 months prior to Screening.

Exclusion Criteria:

1. The participant is participating in another investigational study or has taken any investigational drug within 30 days prior to Day -1.
2. Has donated blood or experienced acute blood loss (including plasmapheresis) of more than 500 mL within 56 days prior to Day -1.
3. Has a history or clinical manifestations of clinically significant metabolic (including Type 2 Diabetes Mellitus, hypercholesterolemia or dyslipidemia but excluding Type 1 Diabetes Mellitus), endocrinologic, hematologic, pulmonary, cardiovascular, gastrointestinal, neurologic, hepatic, renal, urologic, immunologic, glaucoma, or psychiatric disorders, or tendency for urinary retention.
4. Has a known hypersensitivity to TAK-329, any of its excipients, any compound related to TAK-329, or known hypersensitivity to sulfonamides.
5. Has a history of cataract (including traumatic) or glaucoma or has a positive ophthalmic examination with findings suggestive of a cataract within 7 days prior to or at Check in (Day -1) of Period 1.
6. Has a history indicative of proliferative retinopathy or maculopathy and/or severe neuropathy including gastroparesis.
7. Has a history of severe hypoglycemia requiring emergency medical attention less than 6 months prior to Screening or a medical history suggestive of hypoglycemia unawareness less than 1 year prior to Screening.
8. Has a systolic blood pressure ≥145 mm Hg or a diastolic blood pressure ≥90 mm Hg that is confirmed by a repeat measurement taken at least 30 minutes apart at Screening and Check-in (Day -1) of Period 1.
9. Has a history of drug abuse (defined as illicit drug use) or a history of alcohol abuse (defined as regular or daily consumption of more than 4 alcoholic drinks per day) within 2 years prior to Screening.
10. Has an alanine transaminase or aspartate transaminase level of greater than 1.5 x the upper limit of normal at Screening or Check-in (Day -1), active liver disease, active gall bladder disease, or jaundice
11. Has a thyroid stimulating hormone result out of the euthyroid range at Screening.
12. Is on any non-insulin antidiabetic medication (including oral agents such as metformin or pioglitazone or injectables such as pramlintide or exenatide) or inhaled insulin within 90 days prior to Day -1 of Period 1.
13. Has ingested foods or beverages containing grapefruit juice or Seville-type oranges within 14 days prior to Day 1 of Period 1 or any alcohol-or caffeine containing products or medications within 72 hours prior to Day 1 of each treatment period or anticipates an inability to abstain from these substances for the duration of the study.
14. Has used any drug within 28 days prior to Day 1 of Period 1 that may interfere with the interpretation of study results or are known to cause clinically relevant interference with insulin action or glucose utilization.
15. Has a history of cancer that has not been in remission for at least 5 years prior to the first dose of study drug. (This criterion does not include those subjects with basal cell or stage I squamous cell carcinoma of the skin.)
16. Has a history of organ transplant including islet cells transplantation.
17. Has a known history of human immunodeficiency virus or a positive hepatitis B surface antigen and antibody to hepatitis C result at Screening.
18. Has a positive urine screen for drugs or alcohol breathalyzer at Screening or Day -1 of Period 1.
19. Has any other disease or condition including psychiatric conditions at Screening or at Randomization that, in the opinion of the investigator, may adversely affect his or her participation in the study either by being a safety risk to the subject, affecting any of the pharmacokinetic or pharmacodynamic measurements, or making it difficult to successfully manage and follow the subject according to the protocol.
20. Has a history of abdominal surgery (except laparoscopic cholecystectomy or uncomplicated appendectomy), thoracic, or nonperipheral vascular surgery within 6 months prior to Day -1 of Period 1.
21. Has a history or presence of an abnormal electrocardiogram result at Screening or Day -1 of Period 1 that, in the investigator's opinion, is clinically significant.
22. Has used any tobacco within 28 days prior to Day 1 of Period 1 OR has a positive urine cotinine test at Screening, and is unwilling to abstain from these products for the duration of the study.
23. Has poor peripheral venous access.
24. Has had an acute, clinically significant illness within 30 days prior to Day -1, or any other condition or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for the study.
25. The participant is a study site employee, or an immediate family member (ie, spouse, parent, child, or sibling) of a study site employee involved in the conduct of this study.
26. The participant had an acute, clinically significant illness within 30 days prior to Day -1, or any other condition or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for the study.
27. The participant is unable to understand verbal or written English or any other language for which a certified translation of the approved informed consent is available.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
(AUCGIR 0-360): Area Under the Curve of the Glucose Infusion Rate From Time 0 to 360 minutes post dose Pharmacodynamic Parameter. | On Day 1 in Four Treatment Periods.
  (AUCGIR 0-360) is measure of area under the curve of the glucose infusion rate from time 0 to 360 minutes (6 hours) post dose, measured in minutes during the glucose clamp procedure.
GIRmax: Maximum Observed Glucose Infusion Rate Pharmacodynamic Parameter. | On Day 1 in Four Treatment Periods.
  Maximum observed glucose infusion rate (GIRmax) is the peak glucose infusion rate of a drug after administration, obtained directly from the glucose infusion-time curve, measured in minutes during the glucose clamp procedure.
TGIRmax: Time to Reach the Maximum Glucose Infusion Rate (GIRmax) Pharmacodynamic Parameter. | On Day 1 in Four Treatment Periods.
  TGIRmax: Time to reach the maximum Glucose Infusion Rate (GIRmax), equal to time (hours) to GIRmax, measured in minutes during the glucose clamp procedure.

SECONDARY OUTCOMES:
Maximum Observed Pharmacodynamic Response (Emax) of Cortisol During Hypoglycemic Clamp. | On Day 1 in Four Treatment Periods.
  The maximum observed increase or decrease (peak) effect for cortisol, based off sample collected at the start of the clamp procedure, 0 hours predose, and 0. 5, 1.0, 2, 3, 4 and 6 hours postdose. Hypoglycemic clamp procedure is a method for quantifying insulin secretion and resistance, used to measure glucose metabolism and insulin sensitivity.
Area under the effect versus time curves (AUEC) of Cortisol During Hypoglycemic Clamp. | On Day 1 in Four Treatment Periods.
  Area under the effect-time curve calculated using the linear trapezoidal rule for cortisol, based off sample collected at the start of the clamp procedure, 0 hours predose, and 0. 5, 1.0, 2, 3, 4 and 6 hours postdose. Hypoglycemic clamp procedure is a method for quantifying insulin secretion and resistance, used to measure glucose metabolism and insulin sensitivity.
Incidence of Treatment-Emergent Adverse Events. | After receiving first dose of study drug and within 30 days after receiving the last dose of study drug.
  Incidence of treatment-emergent adverse events (TEAE) are adverse events with an onset that occurs after receiving study drug and within 30 days after receiving the last dose of study drug. A TEAE may also be a pretreatment adverse event or a concurrent medical condition diagnosed prior to the date of first dose of study drug that increases in severity after the start of dosing.
Incidence of Hypoglycemia. | After receiving first dose of study drug and Day 7 +/-2 after receiving the last dose of study drug.
  Incidence of hypoglycemia (abnormal low blood sugar) classified into 4 categories: Severe Hypoglycemia (participant experiences confusion or disorientation requiring resuscitative action); Symptomatic Hypoglycemia (blood glucose of <55 mg/dL accompanied by clinically significant signs and symptoms of hypoglycemia); Biochemical Hypoglycemia (blood glucose <50 mg/dL preferably confirmed by second reading, regardless of accompanying symptoms or signs of hypoglycemia); and Other Hypoglycemia (any signs or symptoms considered by investigator indicative of hypoglycemia, regardless of glucose value).

CONTACTS AND LOCATIONS:
Overall Officials: Associate Medical Director, Clinical Science, Study Director — Takeda
Locations (1):
- Chula Vista, California, United States